CLINICAL TRIAL: NCT04572841
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study of the Safety, Tolerability, Pharmacokinetics, and Therapeutic Efficacy of SAR441344 in Adult Patients With Primary Sjögren's Syndrome (pSjS)
Brief Title: Safety, Tolerability, Pharmacokinetics, and Therapeutic Efficacy of SAR441344 in Primary Sjögren's Syndrome (pSjS)
Acronym: phaethuSA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT16618; U1111-1244-2266 (Registry Identifier: ICTRP); 2020-000511-77 (EudraCT Number)
Record Dates: First submitted 2020-09-28; First posted 2020-10-01 (Actual); Results first posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Sjögren's Syndrome; Sjogren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SAR441344 (Experimental): SAR441344 single intravenous (IV) loading dose on Day 1 followed by a single subcutaneous (SC) dose administered once every 2 weeks from Week 2 to Week 10 (5 administrations)
  Interventions: Drug: SAR441344
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAR441344 — Pharmaceutical form: solution for injection
  Route of administration: intravenous or subcutaneous
  Arms: SAR441344
Drug: Placebo — Pharmaceutical form: solution for injection
  Route of administration: intravenous or subcutaneous
  Arms: Placebo

SUMMARY:
Primary Objective:

To evaluate the therapeutic efficacy of one dose level of SAR441344 versus placebo over 12 weeks in adult patients with primary Sjögren's syndrome (pSjS), assessed by the change of the European League Against Rheumatism (EULAR) Sjögren's Syndrome Disease Activity Index (ESSDAI)

Secondary Objectives:

* To evaluate the therapeutic efficacy of one dose level of SAR441344 versus placebo over 12 weeks in adult patients with pSjS
* To evaluate the therapeutic efficacy on fatigue of one dose level of SAR441344 versus placebo over 12 weeks in adult patients with pSjS
* To evaluate the pharmacokinetic (PK) exposure of one dose level of SAR441344 over 12 weeks in adult patients with pSjS
* To evaluate the safety and tolerability of one dose level of SAR441344 versus placebo in adult patients with pSjS as determined by adverse events (AEs)
* To evaluate the local tolerability of one dose level of SAR441344 versus placebo over 12 weeks in adult patients with pSjS
* To evaluate the safety and tolerability of one dose level of SAR441344 versus placebo over 12 weeks in adult patients with pSjS determined by electrocardiogram, vital signs, and laboratory evaluations
* To measure the immunogenicity of one dose level of SAR441344 versus placebo over 12 weeks in adult patients with pSjS

This is a multicenter, randomized, double blind, placebo controlled, parallel group proof of concept Phase 2 study to evaluate the therapeutic efficacy of SAR441344 in adult patients with primary Sjögren's syndrome (pSjS), as well as safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD).

* Study visit frequency: every 2 weeks in the treatment period and every 4 weeks in the follow-up period.
* The total duration of the study will be 24 weeks (28 weeks including maximum screening duration) for each participant, including a 12-week treatment period and a 12-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 80 years of age inclusive, at the time of signing the informed consent.
* Diagnosis of pSjS according to the American College of Rheumatology/EULAR 2016 criteria at Screening.
* Disease duration since first diagnosis of pSjS ≤15 years based on medical history.
* Participants with moderate to severe disease activity set with ESSDAI total score ≥5, based on the following domains at Screening: glandular, articular, muscular, hematological, biological, and constitutional, lymphadenopathy.
* Seropositive for anti-Ro/SSA antibodies.
* IgG > lower limit of normal (ULN) at Screening.
* Stimulated salivary flow rate of ≥0.1 mL/min at Screening or Baseline.
* Body weight within 45 to 120 kg (inclusive) and body mass index within the range of 18.0 to 35.0 kg/m2 (inclusive) at Screening.
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Any autoimmune disease (except pSjS and Hashimoto thyroiditis) with or without secondary SjS.
* History, clinical evidence, suspicion or significant risk for thromboembolic events, as well as myocardial infarction, stroke, and/or antiphospholipid syndrome and any participants requiring antithrombotic treatment.
* Active life threatening or organ threatening complications of pSjS disease at the time of Screening based on treating physician evaluation including but not restricted to:

  * Vasculitis with renal, digestive, cardiac, pulmonary, or CNS involvement characterized as severe,
  * Active central nervous system (CNS) or peripheral nervous system (PNS) involvement requiring high dose steroids,
  * Severe renal involvement defined by objective measures,
  * Lymphoma.
* Cardiac heart failure Stage III or IV according to the New York Heart Association.
* Severe pulmonary impairment documented by an abnormal pulmonary function test.
* Serious systemic viral, bacterial or fungal infection (eg, pneumonia, pyelonephritis), infection requiring hospitalization or IV antibiotics or significant chronic viral (including history of recurrent or active herpes zoster), bacterial, or fungal infection (eg, osteomyelitis) 30 days before and during Screening.
* Participants with a history of invasive opportunistic infections, such as, but not limited to histoplasmosis, listeriosis, coccidioidomycosis, candidiasis, pneumocystis jirovecii, and aspergillosis, regardless of resolution.
* Evidence of active or latent tuberculosis (TB) as documented by medical history (eg, chest X rays) and examination, and TB testing: A positive or 2 indeterminate QuantiFERON® TB Gold tests at Screening (regardless of prior treatment status).
* Evidence of any clinically significant, severe or unstable, acute or chronically progressive, uncontrolled infection or medical condition (eg, cerebral, cardiac, pulmonary, renal, hepatic, gastrointestinal, neurologic, or any known immune deficiency) or previous, active or pending surgical disorder, or any condition that may affect participant safety in the judgment of the Investigator (including vaccinations which are not updated based on local regulation).
* History or presence of diseases which exclude diagnosis of SjS as per the American College of Rheumatology/EULAR 2016 criteria including, but not limited to, sarcoidosis, amyloidosis, graft-versus-host disease, IgG4 related disease, and history of head and neck radiation treatment.
* History of systemic hypersensitivity reaction or significant allergies, other than localized injection site reaction, to any humanized monoclonal antibody.
* Clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe post treatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear IgA dermatosis, toxic epidermal necrolysis, and exfoliative dermatitis).
* Any prior history of malignancy or active malignancy, including lymphoproliferative diseases and lymphoma (except successfully treated carcinoma in situ of the cervix, nonmetastatic squamous cell or basal cell carcinoma of the skin) within 5 years prior to Baseline.
* Unstable dose of nonsteroidal anti inflammatory drugs (NSAIDs) and/or unstable use of topical and/or pharmacological stimulant treatment for salivary and lacrimal glands 4 weeks before Screening.
* High dose steroids, or a change in steroid dose within 4 weeks prior to Day 1/Randomization or expected changes during the course of the study.
* High dose of hydroxychloroquine or chloroquine, or methotrexate or change in hydroxychloroquine, chloroquine or methotrexate dose within 12 weeks prior to Day 1/Randomization or expected changes during the course of the study.
* Participants treated with the following medications/procedures prior to Screening:

  * Previous treatment with azathioprine and other thiopurines, mycophenolate mofetil, sulfasalazine, or cyclosporine A within 3 months.
  * Previous treatment with cyclophosphamide, leflunomide, or belimumab within 6 months.
  * Previous treatment with rituximab within 12 months.
  * Previous bone marrow transplantation, total lymphoid irradiation or ablative ultra high dose cyclophosphamide or IV Ig.
  * Previous treatment with any other biologic drug within 5 times the half life of the drug.
* Received administration of any live (attenuated) vaccine within 3 months prior to Day 1/Randomization (eg, varicella zoster vaccine, oral polio, rabies).
* Clinically significant abnormal ECG or vital signs at Screening.
* Abnormal laboratory test(s) at Screening.
* Positive human immunodeficiency virus (HIV) serology (anti HIV1 and anti HIV2 antibodies) or a known history of HIV infection, active or in remission.
* Positive result on any of the following tests: hepatitis B surface antigen (HBsAg), anti hepatitis B core antibodies (anti HBc Ab), anti hepatitis C virus antibodies (HCV-Ab).
* If female, pregnant and/or breastfeeding.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2024-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (36):
- United States (4):
  - Omega Research Consultants Debary Site Number : 8400005, DeBary, Florida
  - Altoona Center For Clinical Research Site Number : 8400001, Duncansville, Pennsylvania
  - Ramesh C. Gupta, M.D. Site Number : 8400007, Memphis, Tennessee
  - Prolato Clinical Research Center Site Number : 8400009, Houston, Texas
- Argentina (4):
  - Investigational Site Number : 0320004, CABA, Buenos Aires
  - Investigational Site Number : 0320002, CABA, Buenos Aires
  - Investigational Site Number : 0320003, Pergamino, Buenos Aires
  - Investigational Site Number : 0320001, San Miguel de Tucumán, Tucumán Province
- Belgium (2):
  - Investigational Site Number : 0560002, Ghent
  - Investigational Site Number : 0560001, Leuven
- Investigational Site Number : 1240001, Sherbrooke, Quebec, Canada
- Chile (3):
  - Investigational Site Number : 1520002, Osorno, Los Lagos Region
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520004, Viña del Mar, Región de Valparaíso
- France (6):
  - Investigational Site Number : 2500003, Limoges
  - Investigational Site Number : 2500005, Marseille
  - Investigational Site Number : 2500001, Montpellier
  - Investigational Site Number : 2500004, Paris
  - Investigational Site Number : 2500006, Paris
  - Investigational Site Number : 2500002, Strasbourg
- Investigational Site Number : 2760001, Berlin, Germany
- Hungary (3):
  - Investigational Site Number : 3480003, Budapest
  - Investigational Site Number : 3480001, Debrecen
  - Investigational Site Number : 3480004, Székesfehérvár
- Mexico (3):
  - Investigational Site Number : 4840002, Mexicali, Estado de Baja California
  - Investigational Site Number : 4840001, Monterrey, Nuevo León
  - Investigational Site Number : 4840003, Chihuahua City
- South Korea (3):
  - Investigational Site Number : 4100004, Daegu, Daegu
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100001, Seoul
- Spain (2):
  - Investigational Site Number : 7240003, Seville, Andalusia
  - Investigational Site Number : 7240002, Málaga
- Taiwan (4):
  - Investigational Site Number : 1580002, Taichung
  - Investigational Site Number : 1580003, Tainan
  - Investigational Site Number : 1580001, Taipei
  - Investigational Site Number : 1580005, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: ACT16618 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25196&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 35 centers in 12 countries. A total of 234 participants were screened from 12 November 2020 to 10 August 2023, of which 150 were screen failures. Screen failures were mainly due to not meeting the eligibility criteria.
Pre-assignment Details: A total of 84 participants were randomized in a ratio of 1:1 to either placebo or SAR441344 (frexalimab) arm. Randomization was stratified by Baseline European League Against Rheumatism (EULAR) Sjögren's Syndrome Patient Reported Index (ESSPRI) score greater than or equal to (≥) 5 versus less than (<) 5.
Groups:
- Placebo: Participants received a single intravenous (IV) loading dose of placebo matched to SAR441344 on Day 1, followed by a subcutaneous (SC) dose of placebo matched to SAR441344 administered once every 2 weeks (q2w) at Weeks 2, 4, 6, 8 and 10.
- SAR441344: Participants received a single IV loading dose of SAR441344 1200 milligram (mg) on Day 1, followed by an SC dose of SAR441344 600 mg administered q2w at Weeks 2, 4, 6, 8 and 10.
Period: Overall Study
Arm/Group | Placebo | SAR441344
Started | 42 | 42
Completed | 39 | 40
Not Completed | 3 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants exposed to the investigational medicinal product (IMP) (regardless of the amount of treatment administered).
Groups:
- Placebo: Participants received a single IV loading dose of placebo matched to SAR441344 on Day 1, followed by an SC dose of placebo matched to SAR441344 administered q2w at Weeks 2, 4, 6, 8 and 10.
- SAR441344: Participants received a single IV loading dose of SAR441344 1200 mg on Day 1, followed by an SC dose of SAR441344 600 mg administered q2w at Weeks 2, 4, 6, 8 and 10.
- Total: Total of all reporting groups
Arm/Group | Placebo | SAR441344 | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (12.9) | 49.2 (11.1) | 48.5 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 34 | 28 | 62
  Black or African American | 1 | 4 | 5
  Asian | 5 | 4 | 9
  American Indian or Alaska Native | 1 | 6 | 7
  Missing/Not reported | 1 | 0 | 1
EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) Score [Mean (Standard Deviation); unit: score on a scale] — ESSDAI:validated and established outcome measurement for therapeutic efficacy in Sjögren's syndrome, evaluating disease activity mainly on extra-glandular manifestations, and consisted of 12 organ-specific domains(constitutional,lymphadenopathy,glandular,articular,cutaneous,pulmonary, renal,muscular,peripheral and central nervous system,hematological,biological), scored based on organ-specific items in 3 to 4 different severity grades (0=no to 3=high). These scores were summed up in weighted way to summarize into total score ranging from 0-123. Higher scores=worse outcome.
  score on a scale | 10.38 (3.64) | 8.43 (3.88) | 9.40 (3.87)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in ESSDAI Score
Description: ESSDAI is validated and established outcome measurement for therapeutic efficacy in Sjögren's syndrome, evaluating disease activity mainly on extra-glandular manifestations. This score consists of 12 organ-specific domains (constitutional, lymphadenopathy, glandular, articular, cutaneous, pulmonary, renal, muscular, peripheral and central nervous system, hematological, biological), which are scored based on organ-specific items in 3 to 4 different severity grades (no, low, moderate, high; with 0=no and 3=high). These scores are summed up over all 12 domains in weighted way (severity grades are multiplied with weights ranging 1-6 depending on domain) to summarize into total score(0-123). Higher scores indicates worse outcome. Negative change from baseline indicates improvement. Baseline=Day 1 assessment value. Least squares (LS) mean is calculated using mixed models for repeated measures (MMRM). Observed values after occurrence of intercurrent events are excluded.
Time Frame: Baseline (Day 1) to Week 12
Population: Efficacy population included all randomly assigned participants who actually received at least 1 complete dose of IMP with at least 1 post-IMP administration measurement, with available Baseline assessment of the ESSDAI. Only participants with data collected for this outcome measure are reported.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAR441344
Number analyzed (Participants) | 36 | 38
score on a scale | -5.60 (0.60) | -5.29 (0.59)
Statistical Analysis 1: Comparison: Placebo vs SAR441344; Analysis was performed for change from baseline using a mixed model for repeated measures with visit, intervention group (SAR441344 and Placebo), and visit by intervention group interaction as fixed categorical effects, and participant specific baseline ESSDAI as continuous covariate; Test type: Superiority; Least Square Mean Difference = 0.32, 95% CI 2-sided [-1.39 to 2.02], Standard Error of Mean 0.85

2. Secondary Outcome: Change From Baseline to Week 12 in European League Against Rheumatism (EULAR) Sjögren's Syndrome Patient Reported Index (ESSPRI) Score
Description: The ESSPRI is a validated and established outcome measurement, reported by participants, which rates the key disease manifestations: fatigue, dryness, and pain, based on a numeric scale ranging from 0 to 10, where 0 is defined as no symptoms and 10 as maximum imaginable complaints. The total score is the mean score of the 3 scales and ranges from 0 to 10. Higher scores indicates worse outcome. A negative change from baseline indicates improvement. Baseline is defined as Day 1 assessment value. LS mean is calculated using MMRM. Observed values after occurrence of intercurrent events are excluded.
Time Frame: Baseline (Day 1) to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAR441344
Number analyzed (Participants) | 38 | 38
score on a scale | -2.21 (0.34) | -1.92 (0.34)

3. Secondary Outcome: Change From Baseline to Week 12 in Multidimensional Fatigue Inventory (MFI) General Fatigue Subscale and Other Subscales Score
Description: The MFI is a validated, 20 item self-report instrument to evaluate fatigue by investigating the following subscales: general fatigue, physical fatigue, mental fatigue, reduced motivation, and reduced activity. Each subscale consists of 4 items that are scored using a scale from 1 ("yes, this is true") to 5 ("no, this is not true") on which the participants indicate how the listed statements applied to their current fatigue situation. Item scores are summed to create individual subscale score ranging from 4 to 20. A higher score indicates a higher degree of fatigue. A negative change from baseline indicates improvement. Baseline is defined as Day 1 assessment value. LS mean is calculated using ANCOVA. Observed values after occurrence of intercurrent events are excluded.
Time Frame: Baseline (Day 1) to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAR441344
Number analyzed (Participants) | 38 | 38
score on a scale
  General Fatigue Scale Score | 0.37 (0.30) | -0.18 (0.30)
  Mental Fatigue Scale Score | 0.26 (0.36) | 0.37 (0.36)
  Physical Fatigue Scale Score | 0.27 (0.36) | -0.30 (0.36)
  Reduced Activity Scale Score: number analyzed (Participants) | 37 | 38
  Reduced Activity Scale Score | 0.22 (0.31) | 0.29 (0.31)
  Reduced Motivation Scale Score: number analyzed (Participants) | 37 | 38
  Reduced Motivation Scale Score | 0.30 (0.30) | 0.26 (0.29)

4. Secondary Outcome: Mean Plasma Concentration of SAR441344
Description: Blood samples were collected at the specified timepoints for the measurement of plasma concentrations of SAR441344.
Time Frame: At end of infusion and 4 hours post-infusion on Day 1; pre-dose at Weeks 2, 4, 6, 8, 10, and at Week 12
Population: Pharmacokinetic (PK) population included all randomized and treated participants (safety population) with adequate PK results. Participants who received only placebo were not a part of the PK population. Only participants with data collected at specified timepoints for each specified category are reported.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | SAR441344
Number analyzed (Participants) | 39
microgram per milliliter (mcg/mL)
  Day 1 (end of infusion): number analyzed (Participants) | 21
  Day 1 (end of infusion) | 466.10 (93.86)
  Day 1 (4 hours post-infusion): number analyzed (Participants) | 36
  Day 1 (4 hours post-infusion) | 427.22 (102.07)
  Week 2 (pre-dose) | 139.98 (28.30)
  Week 4 (pre-dose) | 132.91 (36.21)
  Week 6 (pre-dose): number analyzed (Participants) | 38
  Week 6 (pre-dose) | 135.18 (46.39)
  Week 8 (pre-dose): number analyzed (Participants) | 38
  Week 8 (pre-dose) | 141.34 (44.85)
  Week 10 (pre-dose): number analyzed (Participants) | 38
  Week 10 (pre-dose) | 142.25 (48.80)
  Week 12: number analyzed (Participants) | 36
  Week 12 | 151.59 (56.49)

5. Secondary Outcome: Median Plasma Concentration of SAR441344
Description: Blood samples were collected at the specified timepoints for the measurement of plasma concentrations of SAR441344.
Time Frame: At end of infusion and 4 hours post-infusion on Day 1; pre-dose at Weeks 2, 4, 6, 8, 10, and at Week 12
Population: PK population included all randomized and treated participants (safety population) with adequate PK results. Participants who received only placebo were not a part of the PK population. Only participants with data collected at specified timepoints for each specified category are reported.
Measure: Median (Full Range); unit: mcg/mL
Arm/Group | SAR441344
Number analyzed (Participants) | 39
mcg/mL
  Day 1 (end of infusion): number analyzed (Participants) | 21
  Day 1 (end of infusion) | 479.06 [302.4 to 652.2]
  Day 1 (4 hours post-infusion): number analyzed (Participants) | 36
  Day 1 (4 hours post-infusion) | 408.37 [253.1 to 623.6]
  Week 2 (pre-dose) | 132.21 [98.3 to 203.1]
  Week 4 (pre-dose) | 133.01 [45.6 to 236.5]
  Week 6 (pre-dose): number analyzed (Participants) | 38
  Week 6 (pre-dose) | 127.32 [60.2 to 237.5]
  Week 8 (pre-dose): number analyzed (Participants) | 38
  Week 8 (pre-dose) | 135.10 [76.9 to 284.9]
  Week 10 (pre-dose): number analyzed (Participants) | 38
  Week 10 (pre-dose) | 134.39 [58.0 to 268.1]
  Week 12: number analyzed (Participants) | 36
  Week 12 | 148.11 [64.4 to 306.2]

6. Secondary Outcome: Maximum Plasma Concentration (Cmax) of SAR441344
Description: Blood samples were collected at the specified timepoints for the measurement of plasma concentrations of SAR441344. Cmax was assessed by a Bayesian approach using the population PK model.
Time Frame: After the last SC dose on Week 10 up to 336 hours post-dose
Population: PK population included all randomized and treated participants (safety population) with adequate PK results. Participants who received only placebo were not a part of the PK population. Only participants with data collected for this outcome measure are reported.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | SAR441344
Number analyzed (Participants) | 38
mcg/mL | 190 (54.5)

7. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of SAR441344
Description: Blood samples were collected at the specified timepoints for the measurement of plasma concentrations of SAR441344. tmax was assessed by a Bayesian approach using the population PK model.
Time Frame: After the last SC dose on Week 10 up to 336 hours post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | SAR441344
Number analyzed (Participants) | 38
hours | 89.1 [76.8 to 139]

8. Secondary Outcome: Area Under the Curve Over the Dosing Interval (AUC0-tau) of SAR441344
Description: Blood samples were collected at the specified timepoints for the measurement of plasma concentrations of SAR441344. AUC0-tau was assessed by a Bayesian approach using the population PK model.
Time Frame: After the last SC dose on Week 10 up to 336 hours post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: microgram*hour per milliliter (mcg*h/mL)
Arm/Group | SAR441344
Number analyzed (Participants) | 38
microgram*hour per milliliter (mcg*h/mL) | 57900 (18000)

9. Secondary Outcome: Terminal Half-life (t1/2z) of SAR441344
Description: Blood samples were collected at the specified timepoints for the measurement of plasma concentrations of SAR441344. t1/2z was assessed by a Bayesian approach using the population PK model.
Time Frame: Week 10 to Week 12
Population: PK population included all randomized and treated participants (safety population) with adequate PK results. Participants who received only placebo were not a part of the PK population.
Measure: Median (Full Range); unit: hours
Arm/Group | SAR441344
Number analyzed (Participants) | 42
hours | 662 [374 to 997]

10. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Treatment-emergent Serious Adverse Events (TESAEs), and Adverse Events of Special Interest (AESI)
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of IMP, whether or not considered related to the IMP. TEAEs: AEs that occurred, worsened, or became serious during the TEAE period (time from the first IMP administration up to Week 24). Serious adverse events (SAE): Any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, or was a congenital anomaly/birth defect. An AESI: an AE (serious or nonserious) of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and immediate notification by the Investigator to the Sponsor was required.
Time Frame: From first dose of IMP (Day 1) up to end of follow-up period (Week 24)
Population: Safety population included all randomized participants exposed to the IMP (regardless of the amount of treatment administered).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAR441344
Number analyzed (Participants) | 42 | 42
Participants
  Any TEAE | 26 | 29
  Any TESAE | 1 | 1
  Any AESI | 5 | 4

11. Secondary Outcome: Number of Participants With Treatment Discontinuation and Withdrawals Due to TEAEs
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of IMP, whether or not considered related to the IMP. TEAEs were AEs that occurred, worsened, or became serious during the TEAE period (time from the first IMP administration up to Week 24).
Time Frame: From first dose of IMP (Day 1) up to end of follow-up period (Week 24)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAR441344
Number analyzed (Participants) | 42 | 42
Participants
  Treatment discontinuation due to TEAEs | 4 | 4
  Treatment withdrawal due to TEAEs | 0 | 0

12. Secondary Outcome: Number of Participants With Increase in Pain Intensity Compared to Pre-dose Pain Intensity at Injection Site by Verbal Descriptor Scale (VDS)
Description: For the measurement of local tolerability, participants had a self-evaluation using a VDS before IMP administration, after completion of the IMP administration, and 2 hours post-administration. The participants were asked to report sensations at the injection site and rated the pain severity as following grading: 0= no pain; 1= mild pain; 2= moderate pain, 3= severe pain, 4= very severe. A positive change in VDS score indicated a higher pain severity compared to the pre-dose pain. The numerical change provides the number of grades the pain got worse (positive change) or improved (negative change). Total number of participants with pain intensity increase (change in VDS score of greater than or equal to 1) compared to pre-dose pain intensity are reported.
Time Frame: Pre-dose (within 24 hours prior IMP dosing), post-dose (up to 15 minutes after dosing) and 2 hours post-dose at Weeks 2, 4, 6, 8 and 10
Population: Safety population included all randomized participants exposed to the IMP (regardless of the amount of treatment administered). Only participants with data collected at specified timepoints for each specified category are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAR441344
Number analyzed (Participants) | 42 | 40
Participants
  Week 2: Post-dose versus pre-dose | 7 | 7
  Week 2: 2 hours post-dose versus pre-dose | 5 | 8
  Week 4: Post-dose versus pre-dose: number analyzed (Participants) | 39 | 40
  Week 4: Post-dose versus pre-dose | 12 | 8
  Week 4: 2 hours post-dose versus pre-dose: number analyzed (Participants) | 39 | 40
  Week 4: 2 hours post-dose versus pre-dose | 5 | 6
  Week 6: Post-dose versus pre-dose: number analyzed (Participants) | 41 | 38
  Week 6: Post-dose versus pre-dose | 13 | 10
  Week 6: 2 hours post-dose versus pre-dose: number analyzed (Participants) | 41 | 38
  Week 6: 2 hours post-dose versus pre-dose | 3 | 3
  Week 8: Post-dose versus pre-dose: number analyzed (Participants) | 39 | 38
  Week 8: Post-dose versus pre-dose | 7 | 11
  Week 8: 2 hours post-dose versus pre-dose: number analyzed (Participants) | 39 | 38
  Week 8: 2 hours post-dose versus pre-dose | 3 | 1
  Week 10: Post-dose versus pre-dose: number analyzed (Participants) | 37 | 38
  Week 10: Post-dose versus pre-dose | 7 | 10
  Week 10: 2 hours post-dose versus pre-dose: number analyzed (Participants) | 37 | 38
  Week 10: 2 hours post-dose versus pre-dose | 5 | 1

13. Secondary Outcome: Number of Participants With AEs Related to Local Tolerability Findings
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of IMP, whether or not considered related to the IMP. Local tolerability at injection site was assessed following IMP injection and findings at the site of injection such as injection site erythema, injection site reaction, and injection site pain were recorded.
Time Frame: Baseline (Day 1) to Week 10
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAR441344
Number analyzed (Participants) | 42 | 42
Participants
  Injection site erythema | 1 | 3
  Injection site reaction | 2 | 0
  Injection site pain | 1 | 0

14. Secondary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities (PCSA) in Vital Signs
Description: PCSA values were defined as abnormal values considered medically important by the Sponsor, according to predefined criteria/thresholds based on literature reviews and defined by the Sponsor. Criteria for PCSA: Sitting systolic blood pressure (SSBP) less than or equal to (≤)95 millimeters of mercury (mmHg) and decrease from baseline ≥20 mmHg; ≥160 mmHg and increase from baseline ≥20 mmHg; Sitting diastolic blood pressure (SDBP) ≤45 mmHg and decrease from baseline ≥10 mmHg, ≥110 mmHg and increase from baseline ≥10 mmHg; Sitting heart rate (HR) ≤50 beats per minute (bpm) and decrease from baseline ≥20 bpm, ≥120 bpm and increase from baseline ≥20 bpm; Weight ≥5% decrease from baseline, ≥5% increase from baseline.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAR441344
Number analyzed (Participants) | 42 | 42
Participants
  SSBP: ≤95 mmHg; decrease from baseline ≥20 mmHg | 2 | 2
  SSBP: ≥160 mmHg; increase from baseline ≥20 mmHg | 0 | 0
  SDBP: ≤45 mmHg; decrease from baseline ≥10 mmHg | 0 | 0
  SDBP: ≥110 mmHg; increase from baseline ≥10 mmHg | 0 | 0
  Sitting HR: ≤50 bpm; decrease from baseline ≥20 bpm | 1 | 0
  Sitting HR: ≥120 bpm; increase from baseline ≥20 bpm | 0 | 0
  Weight: ≥5% decrease from baseline | 6 | 3
  Weight: ≥5% increase from baseline | 2 | 3

15. Secondary Outcome: Number of Participants With PCSA in Electrocardiogram
Description: PCSA values were defined as abnormal values considered medically important by the Sponsor, according to predefined criteria/thresholds based on literature reviews and defined by the Sponsor. Criteria for PCSA: HR <50 bpm, <40 bpm, >90 bpm, >90 bpm and increase from baseline ≥20 bpm, >100 bpm; PR interval, aggregate >200 milliseconds (msec), >200 msec and increase from baseline ≥25%, >220 msec, >220 msec and increase from baseline ≥25%, >240 msec, >240 msec and increase from baseline ≥25%; QRS duration, aggregate >110 msec, >110 msec and increase from baseline ≥25%, >120 msec, >120 msec and increase from baseline ≥25%; QT interval, aggregate >500 msec; corrected QT (QTc) correction method unspecified >450 msec, >480 msec, increase from baseline [30-60] msec, increase from baseline >60 msec.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAR441344
Number analyzed (Participants) | 42 | 42
Participants
  HR: <50 bpm | 2 | 1
  HR: <40 bpm | 0 | 0
  HR: >90 bpm | 3 | 1
  HR: >90 bpm; increase from baseline ≥20 bpm | 1 | 0
  HR: >100 bpm | 0 | 0
  PR interval, aggregate: >200 msec | 4 | 2
  PR interval, aggregate: >200 msec; increase from baseline ≥25% | 1 | 0
  PR interval, aggregate: >220 msec | 1 | 0
  PR interval, aggregate: >220 msec; increase from baseline ≥25% | 0 | 0
  PR interval, aggregate: >240 msec | 1 | 0
  PR interval, aggregate: >240 msec; increase from baseline ≥25% | 0 | 0
  QRS duration, aggregate: >110 msec | 2 | 0
  QRS duration, aggregate: >110 msec; increase from baseline ≥25% | 0 | 0
  QRS duration, aggregate: >120 msec | 1 | 0
  QRS duration, aggregate: >120 msec; increase from baseline ≥25% | 0 | 0
  QT interval, aggregate: >500 msec | 0 | 0
  QTc correction method unspecified: >450 msec | 5 | 2
  QTc correction method unspecified: >480 msec | 0 | 0
  QTc correction method unspecified: Increase from baseline[30-60] msec | 3 | 7
  QTc correction method unspecified: Increase from baseline >60 msec | 0 | 0

16. Secondary Outcome: Number of Participants With PCSA in Hematology Parameters
Description: PCSA values were defined as abnormal values considered medically important by the Sponsor, according to predefined criteria/thresholds based on literature reviews and defined by the Sponsor. Criteria for PCSA: Hemoglobin (Hb) ≤115 grams per liter (g/L) (Male [M]) or ≤95 g/L (Female [F]), ≥185 g/L (M) or ≥165 g/L (F), decrease from baseline ≥20 g/L; Hematocrit ≤0.37 volume per volume (v/v) (M) or ≤0.32 v/v (F), ≥0.55 v/v (M) or ≥0.5 v/v (F); Erythrocytes (red blood cells [RBC]) ≥6 x 10^12 per liter (/L); Platelets <100 x 10^9/L, ≥700 x 10^9/L; Leukocytes (white blood cells [WBC]) <3 x 10^9/L (Non-Black[NB]) or <2 x 10^9/L (Black[B]), ≥16 x 10^9/L; Neutrophils <1.5 x 10^9/L (NB) or <1 x 10^9/L (B); Lymphocytes >4 x 10^9/L, <0.5 x 10^9L; Monocytes >0.7 x 10^9/L; Basophils >0.1 x 10^9/L; Eosinophils >0.5 x 10^9/L or >upper limit of normal(ULN) (if ULN ≥0.5 x 10^9/L).
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAR441344
Number analyzed (Participants) | 42 | 42
Participants
  Hb: ≤115 g/L (M); ≤95 g/L (F) | 0 | 1
  Hb: ≥185 g/L (M); ≥165 g/L (F) | 0 | 1
  Hb: Decrease from baseline ≥20 g/L | 2 | 2
  Hematocrit: ≤0.37 v/v (M); ≤0.32 v/v (F) | 5 | 3
  Hematocrit: ≥0.55 v/v (M); ≥0.5 v/v (F) | 0 | 1
  RBC: ≥6 x 10^12/L | 0 | 1
  Platelets: <100 x 10^9/L | 0 | 0
  Platelets: ≥700 x 10^9/L | 0 | 0
  WBC: <3 x 10^9/L (NB); <2 x 10^9/L (B) | 8 | 5
  WBC: ≥16 x 10^9/L | 0 | 0
  Neutrophils: <1.5 x 10^9/L (NB); <1 x 10^9/L (B) | 7 | 7
  Lymphocytes: >4 x 10^9/L | 0 | 1
  Lymphocytes: <0.5 x 10^9L | 2 | 0
  Monocytes: >0.7 x 10^9/L | 1 | 2
  Basophils: >0.1 x 10^9/L | 0 | 8
  Eosinophils: >0.5 x 10^9/L or >ULN | 1 | 0

17. Secondary Outcome: Number of Participants With PCSA in Clinical Chemistry Parameters
Description: PCSA values:abnormal values considered medically important by Sponsor, according to predefined criteria/thresholds based on literature reviews and defined by Sponsor.Criteria for PCSA:Sodium≤129 millimoles per liter(mmol/L),≥160 mmol/L;Potassium<3 mmol/L,≥5.5 mmol/L;Glucose≤3.9 mmol/L and <lower limit of normal(LLN),≥11.1 mmol/L(unfasted);≥7 mmol/L(fasted); Creatine kinase(CK)>3 ULN,>10 ULN;Creatinine≥150 micromoles/L(adults),≥30% change from baseline,≥100% change from baseline;Creatinine clearance(CG)≥60-<90 milliliters per minute(mL/min)(mild decrease in glomerular filtration rate[GFR]),≥30-<60 mL/min(moderate decrease in GFR),≥15-<30 mL/min(severe decrease in GFR),<15 mL/min(end stage renal disease),Urea nitrogen≥17 mmol/L;Alkaline phosphatase(ALP)>1.5 ULN;Alanine aminotransferase(ALT)>3 ULN; ALT>3 ULN and bilirubin>2 ULN;Aspartate aminotransferase(AST)>3 ULN;Direct bilirubin>35% bilirubin and bilirubin>1.5 ULN;Total bilirubin>1.5 ULN,>2 ULN.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAR441344
Number analyzed (Participants) | 42 | 42
Participants
  Sodium: ≤129 mmol/L | 0 | 0
  Sodium: ≥160 mmol/L | 0 | 0
  Potassium: <3 mmol/L | 0 | 0
  Potassium: ≥5.5 mmol/L | 1 | 0
  Glucose: ≤3.9 mmol/L and <LLN | 3 | 5
  Glucose: ≥11.1 mmol/L (unfasted); ≥7 mmol/L (fasted) | 3 | 1
  CK: >3 ULN | 0 | 1
  CK: >10 ULN | 0 | 0
  Creatinine: ≥150 micromoles/L (Adults) | 0 | 0
  Creatinine: ≥30% change from baseline | 1 | 2
  Creatinine: ≥100% change from baseline | 0 | 0
  CG: ≥60 - <90 mL/min | 24 | 16
  CG: ≥30 - <60 mL/min | 3 | 2
  CG: ≥15 - <30 mL/min | 0 | 0
  CG: <15 mL/min | 0 | 0
  Urea Nitrogen: ≥17 mmol/L | 0 | 0
  ALP: >1.5 ULN | 0 | 1
  ALT: >3 ULN | 0 | 0
  ALT >3 ULN; Bilirubin >2 ULN | 0 | 0
  AST: >3 ULN | 0 | 0
  Direct Bilirubin >35% Bilirubin; Bilirubin >1.5 ULN | 0 | 0
  Total Bilirubin: >1.5 ULN | 0 | 1
  Total Bilirubin: >2 ULN | 0 | 0

18. Secondary Outcome: Number of Participants With PCSA in Urinalysis Parameters
Description: PCSA values were defined as abnormal values considered medically important by the Sponsor, according to predefined criteria/thresholds based on literature reviews and defined by the Sponsor. Criteria for PCSA: Potential of hydrogen (pH) ≤4.6 or ≥8.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAR441344
Number analyzed (Participants) | 42 | 42
Participants
  pH ≤4.6 | 0 | 0
  pH ≥8 | 3 | 2

19. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) to SAR441344
Description: Serum samples were collected at the specified timepoints for the assessment of ADAs to SAR441344. Number of participants with treatment-emergent ADA defined as at least 1 treatment-induced/boosted ADA during the treatment-emergent period, i.e. from the time of the IMP administration up to the end of study visit are reported. Number of participants with positive ADA are reported.
Time Frame: Baseline, Week 4, Week 8, Week 12, and Week 24
Population: ADA population included all randomized participants treated with SAR441344 with at least 1 post-baseline ADA result (positive, negative or inconclusive). Only participants with data collected at specified timepoints are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | SAR441344
Number analyzed (Participants) | 42
Participants
  Baseline | 2
  Week 4: number analyzed (Participants) | 41
  Week 4 | 2
  Week 8: number analyzed (Participants) | 38
  Week 8 | 2
  Week 12 | 0
  Week 24: number analyzed (Participants) | 41
  Week 24 | 5

ADVERSE EVENTS:
Time Frame: From first dose of IMP (Day 1) up to end of follow-up period (Week 24)
Description: Analysis was performed on safety population.
Arm/Group | Placebo | SAR441344
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 1/42 | 1/42
Other Adverse Events (participants affected / at risk) | 20/42 | 15/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=42) | SAR441344 (N=42)
Osteomyelitis Acute (Infections and infestations) | 1 (1) | 0 (0)
Device Breakage (Product Issues) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=42) | SAR441344 (N=42)
Covid-19 (Infections and infestations) | 4 (4) | 4 (4)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 6 (6) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 0 (0) | 3 (4)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Injection Site Erythema (General disorders) | 1 (3) | 3 (7)
Accidental Overdose (Injury, poisoning and procedural complications) | 5 (5) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/41/NCT04572841/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-24): https://cdn.clinicaltrials.gov/large-docs/41/NCT04572841/SAP_001.pdf